CLINICAL TRIAL: NCT03466411
Title: A Phase 2/3, Randomized, Double-blind, Placebo- and Active-controlled, Parallel-group, Multicenter Protocol to Evaluate the Efficacy and Safety of Guselkumab in Participants With Moderately to Severely Active Crohn's Disease
Brief Title: A Study of the Efficacy and Safety of Guselkumab in Participants With Moderately to Severely Active Crohn's Disease
Acronym: GALAXI
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108387; CNTO1959CRD3001 (Other: Janssen Research & Development, LLC); 2017-002195-13 (EudraCT Number); 2023-504736-18-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2018-03-08; First posted 2018-03-15 (Actual); Results first posted 2025-05-07 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — guselkumab; Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Phase 2 (GALAXI 1): Group 1 (Guselkumab) (Experimental): Participants will receive guselkumab (Dose 1) by intravenous (IV) infusion, followed by guselkumab (Dose 2) by subcutaneous (SC) injection. Participants who are eligible and willing to continue guselkumab may enter the Long-Term Extension (LTE) phase and continue to receive guselkumab.
  Interventions: Drug: Guselkumab Dose 1; Drug: Guselkumab Dose 2
- Phase 2 (GALAXI 1): Group 2 (Guselkumab) (Experimental): Participants will receive guselkumab (Dose 3) by intravenous (IV) infusion, followed by guselkumab (Dose 2) by subcutaneous (SC) injection. Participants who are eligible and willing to continue guselkumab may enter the LTE phase and continue to receive guselkumab.
  Interventions: Drug: Guselkumab Dose 2; Drug: Guselkumab Dose 3
- Phase 2 (GALAXI 1): Group 3 (Guselkumab) (Experimental): Participants will receive guselkumab (Dose 4) by intravenous (IV) infusion, followed by guselkumab (Dose 5) by subcutaneous (SC) injection. Participants who are eligible and willing to continue guselkumab may enter the LTE phase and continue to receive guselkumab.
  Interventions: Drug: Guselkumab Dose 4; Drug: Guselkumab Dose 5
- Phase 2 (GALAXI 1): Group 4 (Ustekinumab) (Active Comparator): Participants will receive ustekinumab by intravenous (IV) infusion, followed by subcutaneous (SC) injection. Participants who are eligible and willing to continue ustekinumab may enter the LTE and continue to receive ustekinumab.
  Interventions: Drug: Ustekinumab
- Phase 2 (GALAXI 1): Group 5 (Placebo/Ustekinumab) (Experimental): Participants will receive placebo administered by intravenous (IV) infusion. At Week 12, non-responders will receive active treatment (Ustekinumab) administered by intravenous (IV) infusion followed by subcutaneous (SC) injection. Participants who are eligible and willing to continue placebo/ustekinumab may enter the LTE and continue to receive placebo/ustekinumab.
  Interventions: Drug: Ustekinumab; Drug: Placebo
- Phase 3 (GALAXI 2 and 3): Group 1 and Group 2 (Guselkumab) (Experimental): Participants will receive guselkumab by intravenous (IV) infusion, followed by guselkumab by subcutaneous (SC) injection. Participants who are eligible and willing to continue guselkumab may enter the LTE phase and continue to receive guselkumab.
  Interventions: Drug: Guselkumab
- Phase 3 (GALAXI 2 and 3): Group 3 (Ustekinumab) (Active Comparator): Participants will receive ustekinumab by intravenous (IV) infusion, followed by subcutaneous (SC) injection. Participants who are eligible and willing to continue ustekinumab may enter the LTE phase and continue to receive ustekinumab.
  Interventions: Drug: Ustekinumab
- Phase 3 (GALAXI 2 and 3): Group 4 (Placebo/Ustekinumab) (Experimental): Participants will receive placebo administered by intravenous (IV) infusion. At Week 12, non-responders will receive active treatment (ustekinumab) administered by intravenous (IV) infusion followed by subcutaneous (SC) injection. Participants who are eligible and willing to continue placebo/ustekinumab may enter the LTE and continue to receive placebo/ustekinumab.
  Interventions: Drug: Ustekinumab; Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab Dose 1 — Guselkumab will be administered by IV infusion.
  Arms: Phase 2 (GALAXI 1): Group 1 (Guselkumab)
Drug: Guselkumab Dose 2 — Guselkumab will be administered by SC injection.
  Arms: Phase 2 (GALAXI 1): Group 1 (Guselkumab); Phase 2 (GALAXI 1): Group 2 (Guselkumab)
Drug: Guselkumab Dose 3 — Guselkumab will be administered by IV infusion.
  Arms: Phase 2 (GALAXI 1): Group 2 (Guselkumab)
Drug: Guselkumab Dose 4 — Guselkumab will be administered by IV infusion.
  Arms: Phase 2 (GALAXI 1): Group 3 (Guselkumab)
Drug: Guselkumab Dose 5 — Guselkumab will be by SC injection.
  Arms: Phase 2 (GALAXI 1): Group 3 (Guselkumab)
Drug: Guselkumab — Guselkumab will be administered by IV infusion and SC injection.
  Arms: Phase 3 (GALAXI 2 and 3): Group 1 and Group 2 (Guselkumab)
Drug: Ustekinumab — Ustekinumab will be administered by IV infusion and SC injection.
  Arms: Phase 2 (GALAXI 1): Group 4 (Ustekinumab); Phase 2 (GALAXI 1): Group 5 (Placebo/Ustekinumab); Phase 3 (GALAXI 2 and 3): Group 3 (Ustekinumab); Phase 3 (GALAXI 2 and 3): Group 4 (Placebo/Ustekinumab)
Drug: Placebo — Placebo will be administered as IV infusion.
  Arms: Phase 2 (GALAXI 1): Group 5 (Placebo/Ustekinumab); Phase 3 (GALAXI 2 and 3): Group 4 (Placebo/Ustekinumab)

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy (GALAXI 1), clinical and endoscopic efficacy (GALAXI 2 and GALAXI 3) and safety of guselkumab in participants with Crohn's disease.

DETAILED DESCRIPTION:
This program consists of 3 separate studies: a 48-week Phase 2 dose-ranging study (GALAXI 1) and two 48-week Phase 3 confirmatory studies (GALAXI 2 and GALAXI 3). In Phase 2, safety and efficacy of guselkumab dose regimens will be evaluated to support the selection of induction and maintenance dose regimens for confirmatory evaluation in Phase 3. Participants who complete the 48-week Phase 2 or Phase 3 studies may be eligible to enter the long term extension (LTE). Throughout the 3 studies, efficacy, pharmacokinetic, biomarkers, and safety will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Have Crohn's disease (CD) or fistulizing Crohn's disease of at least 3 months duration (defined as a minimum of 12 weeks), with colitis, ileitis, or ileocolitis, confirmed at any time in the past by radiography, histology, and/or endoscopy
* Have moderate to severe CD as assessed by CDAI, stool frequency (SF), and abdominal pain (AP) scores, and Simple Endoscopic Score for Crohn's Disease (SES-CD)
* Have screening laboratory test results within the protocol specified parameters
* A female participant of childbearing potential must have a negative urine pregnancy test result at screening and baseline
* Demonstrated intolerance or inadequate response to conventional or to biologic therapy for CD

Exclusion Criteria:

* Current diagnosis of ulcerative colitis or indeterminate colitis
* Has complications of Crohn's disease, such as symptomatic strictures or stenoses, short gut syndrome, or any other manifestation
* Unstable doses of concomitant Crohn's disease therapy
* Receipt of Crohn's disease approved biologic agents, investigational agents, or procedures outside of permitted timeframe as specified in the protocol
* Any medical contraindications preventing study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1409 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2028-01-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (575):
- United States (109):
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Internal Medicine Center, Mobile, Alabama
  - University of Arizona, Tucson, Arizona
  - Advanced Research Center Inc, Anaheim, California
  - Paul Wallace MD, Beverly Hills, California
  - University Of California San Diego, La Jolla, California
  - Om Research LLC, Lancaster, California
  - Allameh Medical Corp, Mission Viejo, California
  - United Gastroenterologists, Murrieta, California
  - Clinnova Research, Orange, California
  - Inland Empire Liver Foundation, Rialto, California
  - UC Davis Medical Center, Sacramento, California
  - Clinical Applications Laboratories, Inc, San Diego, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Pioneer Research Solutions Inc., Coconut Creek, Florida
  - InvesClinic, LLC, Fort Lauderdale, Florida
  - Harmony Medical Research Institute, Inc., Hialeah, Florida
  - Elite Research Network - Nature Coast Clinical Research, LLC, Inverness, Florida
  - SIH Research, Kissimmee, Florida
  - Auzmer Research, Lakeland, Florida
  - Florida Research Center Inc., Lakewood Rch, Florida
  - Homestead Associates in Research Inc, Miami, Florida
  - Community Research Foundation, Inc., Miami, Florida
  - Sanchez Clinical Research, Inc, Miami, Florida
  - Visionary Investigators Network, Miami, Florida
  - Gastroenterology Group Of Naples, Naples, Florida
  - Florida Hospital, Orlando, Florida
  - Omega Research Consultants, Orlando, Florida
  - Care Access Research, Orlando, Orlando, Florida
  - Synexus Clinical Research US Inc, Pinellas Park, Florida
  - Central Florida Internists, Saint Cloud, Florida
  - Synergy Clinical Research, St. Petersburg, Florida
  - Theia Clincial Research, LLC, St. Petersburg, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - GCP Clinical Research, Tampa, Florida
  - Florida Hospital Tampa, Tampa, Florida
  - Alliance Clinical Research, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Morehouse School of Medicine, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Atlanta Center For Gastroenterology, Decatur, Georgia
  - Gastroenterology Consultants, Roswell, Georgia
  - Atlanta Gastroenterology Specialists PC, Suwanee, Georgia
  - Carle Foundation Hospital, Urbana, Illinois
  - IU Health University Hospital, Indianapolis, Indiana
  - BVL Clinical Research, Leawood, Kansas
  - Health Science Research Center, Pratt, Kansas
  - Cotton O'Neil Digestive Health Center, Topeka, Kansas
  - Gastroenterology Associates, Baton Rouge, Louisiana
  - Gastroenterology Clinic of Acadiana, Lafayette, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - LSUHSC Shreveport Feist-Weiller Cancer Center, Shreveport, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Woodholme Gastroenterology Associates, Baltimore, Maryland
  - Digestive Health Specialists PC, Chelmsford, Massachusetts
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Huron Gastroenterology Associates Center for Digestive Care, Ypsilanti, Michigan
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Atlantic Digestive Health Institute/ Atlantic IBD Center, Morristown, New Jersey
  - A1 Clinical Research, Jackson Heights, New York
  - Weill Cornell Medical College, New York, New York
  - New York Gastroenterology Associates, New York, New York
  - Care Access Research, New York, New York
  - NYU Langone Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Syracuse VA Medical Center, Syracuse, New York
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - University North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Charlotte Gastroenterology and Hepatology, PLLC, Charlotte, North Carolina
  - Onsite Clinical Solutions, Charlotte, North Carolina
  - Cumberland Research Associates, Fayetteville, North Carolina
  - Care Access Research, Kinston, Kinston, North Carolina
  - Clinical Trials of America, Mount Airy, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Clinical Inquest Center, LTD, Beavercreek, Ohio
  - Ohio State University, Columbus, Ohio
  - Synexus Clinical Research US Inc, Columbus, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Southwoods Health, Poland, Ohio
  - Northshore Gastroenterology Research, LLC, Westlake, Ohio
  - Integris Baptist Office, Oklahoma City, Oklahoma
  - US Digestive Health, Wyomissing, Pennsylvania
  - Synexus Clinical Research US Inc, Anderson, South Carolina
  - Gastroenterology Associates P.A., Greenville, South Carolina
  - Memorial Health Care System, Chattanooga, Tennessee
  - Gastro One, Germantown, Tennessee
  - Tennessee State University, Johnson, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - DHAT Research Institute, Garland, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Houston Digestive Diseases Consultants, Houston, Texas
  - CliniCore Houston, Houston, Texas
  - Caprock Gastro Research, Lubbock, Texas
  - Gastroenterology Clinic Of San Antonio P A, San Antonio, Texas
  - Gastroenterology Research of America, LLC, San Antonio, Texas
  - UT Health Science Center at San Antonio, San Antonio, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Texas Gastroenterology Associates - Research, Spring, Texas
  - Baylor Scott and White Research Institute, Temple, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Center for Gastrointestinal Health, Petersburg, Virginia
  - Gastroenterology Consultants of Southwest Virginia, Roanoke, Virginia
  - Northwest Gastroenterology Associates - USA, Bellevue, Washington
  - Washington Gastroenterology, PLLC, Tacoma, Washington
- Australia (11):
  - The Queen Elizabeth Hospital, Adelaide
  - Monash Health, Monash Medical Centre, Clayton
  - Concord Hospital, Concord
  - Austin Hospital, Heidelberg
  - Sir Charles Gairdner Hospital, Nedlands
  - Royal Adelaide Hospital, North Terrace
  - Royal Melbourne Hospital, Parkville
  - Nepean Hospital, Penrith
  - The Alfred Hospital, Prahran
  - Mater Hospital Brisbane, South Brisbane
  - Princess Alexandra Hospital, Woolloongabba
- Austria (2):
  - Universitaetsklinikum Salzburg Landeskrankenhaus, Salzburg
  - Akh Wien, Vienna
- Belarus (5):
  - Grodno University Hospital, Grodno
  - Gomel Regional Clinical Hospital, Homyel
  - Republican Research Centre of Radiation Medicine and Human E, Homyel
  - Healthcare Institution,Minsk Scientific center for surgery,, Minsk
  - Vitebsk Regional Clinical Hospital, Vitebsk
- Belgium (7):
  - AZ Klina, Brasschaat
  - CHU Saint-Pierre, Brussels
  - Hopital Erasme, Brussels
  - UZ Gent, Ghent
  - Az Groeninge, Kortrijk
  - Algemeen Ziekenhuis Delta, Roeselare
  - CHwapi, Tournai
- Bosnia and Herzegovina (5):
  - University Clinical Centre of the Republic of Srpska, Banja Luka
  - Clinical hospital Mostar, Mostar
  - Clinical Center University of Sarajevo, Sarajevo
  - Polyclinic Dr. Al-Tawil, Sarajevo
  - Cantonal Hospital Zenica, Zenica
- Brazil (24):
  - MK Blumenau Pesquisa Clínica, Blumenau
  - Universidade Estadual Paulista 'Julio De Mesquita Filho', Botucatu
  - L2IP Instituto de Pesquisas Clinicas, Brasília
  - Sociedade Campineira de Educacao e Instrucao Hospital e Maternidade Celso Pierro, Campinas
  - Hospital Nossa Senhora Das Gracas, Curitiba
  - Inst Goiano Gastroenterologia e Endoscopia Digest Ltda - Clinica de Gastro, Goiânia
  - Centro de Estudos Clínicos do Interior Paulista - CECIP, Jaú
  - CMIP - Centro Mineiro de Pesquisa Ltda, Juiz de Fora
  - Complexo Hospitalar de Niteroi, Niterói
  - Instituto Mederi de Pesquisa e Saude, Passo Fundo
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Instituto do Aparelho Digestivo, Porto Alegre
  - Universidade Federal do Rio de Janeiro - Faculdade de Medicina, Rio de Janeiro
  - Hospital Santa Izabel, Salvador
  - Pesquisare Saude, Santo André
  - Praxis pesquisa médica, Santo André
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, Santo André
  - Irmandade da Santa Casa da Misericórdia de Santos, Santos São Paulo
  - Kaiser Hospta, São José do Rio Preto
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
  - CPCLIN - Centro de Pesquisas Clínicas, São Paulo
  - Hemomed, São Paulo
  - BR Trials, São Paulo
  - Fundacao Universidade Federal do Piaui - Universidade Federal do Piaui, Teresina
- Canada (11):
  - University of Calgary, Calgary, Alberta
  - Gastroenterology and Internal Medicine Research Institute (GIRI), Edmonton, Alberta
  - University of Alberta- Ziedler Ledcor Centre, Edmonton, Alberta
  - Columbia Gastroenterology, New Westminster, British Columbia
  - Health Sciences Centre, Winnipeg, Manitoba
  - Barrie GI Associates, Barrie, Ontario
  - London Health Sciences Centre, London, Ontario
  - Mount Sinai Hospital-Toronto, Toronto, Ontario
  - Pharmaceutical Integrated Research Company, Waterloo, Ontario
  - MUHC Montreal General Hospital, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- China (35):
  - Peking University First Hospital, Beijing
  - Beijing Friendship Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The Military General Hospital of Beijing PLA, Beijing
  - The second Xiangya Hospital of Central South University, Changsha
  - Changzhou No 2 Peoples Hospital, Changzhou
  - West China Hospital Sichuan University, Chengdu
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - First Affiliated Hospital of Gannan Medical University, Ganzhou
  - The First Affiliated Hospital Sun Yat-Sen University, Guangzhou
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou
  - ZhuJiang Hospital of Southern Medical University, Guangzhou
  - Sun Yat-sen University - The Sixth Affiliated Hospital Guangdong Gastrointestinal Hospital, Guangzhou
  - The Second Affiliated Hospital of Zhejiang University, Hangzhou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Huai'an 1st Hospital, Huai'an
  - The First Affiliated Hospital of NanChang University, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - Shanghai Ninth Peoples Hospital, Shanghai
  - Huashan Hospital Fudan University, Shanghai
  - Second Military Medical University (SMMU), Shanghai
  - Tongji Hospital of Tongji University, Shanghai
  - Ruijin Hospital Shanghai Jiao Tong University, Shanghai
  - Shengjing Hospital Of China Medical University, Shenyang
  - Peking University Shenzhen Hospital, Shenzhen
  - The first affiliated hospital of suzhou University, Suzhou
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Wuhan Union Hospital, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - Wuxi People s Hospital, Wuxi
  - Zhongshan Hospital, Xiamen University, Xiamen
  - Yangzhou First People's Hospital, Yangzhou
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou
- Colombia (5):
  - Medplus Medicina Prepagada S.A., Bogotá
  - Clinica de la Mujer, Bogotá
  - Endocare Ltda., Bogotá
  - Centro Médico Imbanaco, Cali
  - Corporacion para Estudios en Salud Clinica CES - Gastroenterology, Medellín
- Croatia (6):
  - Opca bolnica Bjelovar, Bjelovar
  - Opca bolnica Zadar, Zadar
  - CH Sestre Milosrdnice, Zagreb
  - Poliklinika Solmed, Zagreb
  - University Hospital Center Zagreb, Zagreb
  - University Hospital Dubrava, Zagreb
- Czechia (6):
  - Nemocnice Ceske Budejovice, České Budějovice
  - NH Hospital, a.s., Hořovice
  - Hepato-gastroenterologie HK, s.r.o., Hradec Králové
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Synexus Czech s.r.o., Prague
  - ISCARE a.s., Prague
- France (23):
  - CHU Amiens, Amiens
  - Centre Hospitalier de la Cote Basque, Bayonne
  - CHRU Besancon Hopital Jean Minjoz, Besançon
  - Centre Hospitalier Universitaire (CHU) de Caen, Caen
  - CHRU de Tours - Hopital Trousseau, Chambray Les Tours Centre
  - Centre Hospitalier Universitaire(CHU) - Hopital Henri Mondor, Créteil
  - CHU Grenoble, Grenoble
  - CHRU de Lille Hopital Claude Huriez, Lille
  - Hopital Nord Marseille, Marseille
  - CHRU Montpellier - Hopital Saint-Eloi, Montpellier
  - CHU de Nantes hotel Dieu, Nantes
  - CHU de Nice Hopital de l Archet, Nice
  - CHU Nimes Hopital Caremeau, Nîmes
  - Hôpital Bichat, Paris
  - Groupement Hospitalier Universitaire Ouest, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Reims, Hôpital Robert Debré, Reims
  - CHU Saint Etienne, Saint-Etienne
  - Hopital D'Instruction Des Armees, Saint-Mandé
  - CHRU de Strasbourg - Hopital de Hautepierre, Strasbourg
  - CHU Toulouse - Hopital de Rangueil, Toulouse
  - Hopital Rangueil, Toulouse
  - CHU de Nancy_ Hopital Brabois, Vandœuvre-lès-Nancy
- Georgia (6):
  - TSMU The First University Clinic, Tbilisi
  - Institute of Clinical Cardiology, Ltd., Tbilisi
  - LTD 'Georgia Archangel St. Michael Multiprofile Clinical Hospital', Tbilisi
  - LTD 'Aversi Clinic', Tbilisi
  - LTD Helsicore, Tbilisi
  - LTD Unimed Kakheti- Telavi Referral Hospital, Telavi
- Germany (23):
  - Klinikum Augsburg, Augsburg
  - Charite - Campus Mitte, Berlin
  - Synexus Berlin Research Center, Berlin
  - Universitaetsklinikum Charite, Campus Virchow Klinikum, Berlin
  - Krankenhaus Waldfriede Mitte, Berlin
  - Klinikum Dresden, Dresden
  - Synexus Clinical Research GmbH, Frankfurt
  - JWG-University Hospital, Frankfurt
  - Agaplesion Frankfurter Diakonie Kliniken GmbH, Markus Krankenhaus, Frankfurt am Main
  - Martini-Klinik am Universitätsklinikum Hamburg-Eppendorf Urologie, Hamburg
  - Asklepios Westklinikum, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Gastroenterologische Spezialpraxis - Berlin-Karlshorst, Karlshorst
  - Universitatsklinikum Schleswig Holstein Kiel, Kiel
  - Eugastro GmbH, Leipzig
  - Gastroenterologie und Hepatologie am Johannisplatz, Leipzig
  - Staedtisches Klinikum Lueneburg, Lüneburg
  - Universitaetsklinikum Mannheim, Mannheim
  - Gemeinschaftspraxis Germania-Campus, Münster
  - Praxiszentrum Alte Mälzerei, Regensburg
  - Zentrum für Gastroenterologie Saar MVZ GmbH, Saarbrücken
  - Universitatsklinikum Ulm, Ulm
- Greece (2):
  - Laiko General Hospital of Athens, Athens
  - University Hospital of Heraklion, Heraklion
- Hungary (7):
  - Réthy Pál Kórház - Rendelőintézet, Békéscsaba
  - Synexus Magyarorszag Kft, Budapest
  - Péterfy Sándor utcai Kórház, Budapest
  - Meddica Centre Hungarian Defence Froces, Budapest
  - Semmelweis Egyetem, Budapest
  - Synexus Magyarorszag Kft, Gyula
  - Tolna Megyei Balassa Janos Korhaz, Szekszárd
- India (8):
  - Apex Hospitals Ltd, Jaipur
  - Fortis Hospital, New Delhi
  - Fortis Hospital, Noida
  - Shree Giriraj Multispeciality Hospital, Rajkot
  - Nirmal Hospital Pvt. Ltd., Surat
  - Surat Institute of Digestive Sciences Hospitals, Surat
  - BAPS Pramukhswami Hospital, Surat
  - Unity Hospital, Surat
- Israel (12):
  - Ha'Emek Medical Center, Afula
  - Barzilai Medical Center, Ashkelon
  - Soroka Medical Center, Bear Sheva
  - Rambam Medical Center, Haifa
  - Bnai Zion Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Hebrew University Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Med Ctr Beilinson Hosp, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assaf Harofeh Medical Center, Tzrifin
- Italy (14):
  - Policlinico S.Orsola Malpighi, AOU di Bologna, Bologna
  - Azienda Ospedaliero Universitaria di Cagliari - Policlinico Duilio Casula di Monserrato, Cagliari
  - Ospedale Santissima Annunziata, Cento
  - AOU Policlinico G.Martino, Messina
  - Gruppo Ospedaliero San Donato - Istituto di Ricovero e Cura, Milan
  - Universita degli Studi di Padova - Azienda Ospedaliera di Padova, Padua
  - Università Campus Biomedico di Roma, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
  - Complesso Integrato Columbus, Rome
  - IRCCS Humanitas Rozzano-IBD Center Malattie Infiammatorie Croniche Intestinali, Rozzano
  - Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - S.C. Gastroenterologia, Torino
  - Azienda Ospedaliero Universitaria S.Maria Della Misericordia, Udine
  - Policlinico G.B.Rossi, Verona
- Japan (76):
  - Asahikawa City Hospital, Asahikawa
  - Tokyo Medical and Dental University Hospital, Bunkyō City
  - Juntendo University Hospital, Bunkyō City
  - Chiba University Hospital, Chiba
  - Fukuoka University Chikushi Hospital, Chikushino-shi
  - Saiseikai Fukuoka General Hospital, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - Gifu University Hospital, Gifu
  - Tokai University Hachioji Hospital, Hachiōji
  - Matsuda Hospital, Hamamatsu
  - Mito Medical Center - Digestive Organs, Higashiibaraki-gun
  - National Hospital Organization Hirosaki General Medical Center, Hirosaki
  - Hiroshima University Hospital, Hiroshima
  - National Hospital Organization Kanazawa Medical Center, Ishikawa
  - Izumiotsu Municipal Hospital, Izumiōtsu
  - Shimane University Hospital, Izumo
  - Kagoshima IBD Gastroenterology Clinic, Kagoshima
  - Sameshima Hospital, Kagoshima
  - Nanpuh Hospital, Kagoshima
  - Kanazawa University Hospital, Kanazawa
  - Nara Medical University Hospital, Kashihara
  - Tsujinaka Hospital Kashiwanoha, Kashiwa
  - The Jikei University Hospital, Kashiwa
  - Aoyama Naika Clinic, Kobe
  - Kobe University Hospital, Kobe
  - National Hospital Organization Kochi National Hospital, Kochi
  - Yamanashi Prefectural Central Hospital, Kofu
  - National Hospital Organization Kure Medical Center and Chugoku Cancer Center, Kure
  - Kurume University Hospital, Kurume
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - JRC Kyoto Daiichi Hospital, Kyoto
  - Kyoto University Hospital, Kyoto
  - National Hospital Organization Kyoto Medical Center, Kyoto
  - Kitasato University Kitasato Institute Hospital, Minatoku
  - Kyorin University Hospital, Mitaka
  - Iwate Medical University Hospital, Morioka
  - Aichi Medical University Hospital, Nagakute
  - Nagaoka Red Cross Hospital, Nagaoka
  - Nagasaki University Hospital, Nagasaki
  - Nagoya University Hospital, Nagoya
  - Nagoya City University Hospital, Nagoya
  - The Hospital of Hyogo College of Medicine, Nishinomiya
  - JA Obihiro Kosei Hospital, Obihiro
  - Okayama Saiseikai General Hospital, Okayama
  - Nakagami Hospital, Okinawa
  - Kinshukai Infusion Clinic, Osaka
  - Kitano Hospital, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka
  - Japanese Red Cross Osaka Hospital, Osaka
  - Osaka City University Hospital, Osaka
  - Oita Red Cross Hospital, Ōita
  - Kindai University Hospital, Ōsaka-sayama
  - Osaki Citizen Hospital, Ōsaki
  - Shiga University of Medical Science Hospital, Ōtsu
  - National Hospital Organization Higashi Ohmi General Medical Center, Ōtsu
  - Japan Community Health Care Organization Saitama Medical Center, Saitama
  - Tokitokai Tokito Clinic Coloproctology Center, Saitama
  - Saitama Medical University Hospital, Saitama
  - Toho University Sakura Medical Center, Sakura
  - JA Sapporo-Kosei General Hospital - 1st Digestive Organs, Sapporo
  - Hokkaido University Hospital, Sapporo
  - Sapporo Higashi Tokushukai Hospital, Sapporo
  - Sapporo IBD Clinic, Sapporo Chuo-ku
  - Tokyo Yamate Medical Center, Shinjuku-ku
  - Osaka University Hospital, Suita-shi
  - Takamatsu Red Cross Hospital, Takamatsu
  - Kagawa Prefectural Central Hospital, Takamatsu
  - Tokushima University Hospital, Tokushima
  - The Jikei University Hospital, Tokyo
  - Yuaikai Tomishiro Central Hospital, Tomishiro
  - Toyama City Hospital, Toyama
  - Fujita Health University Hospital, Toyoake
  - Ehime University Hospital, Tōon
  - Mie University Hospital, Tsu
  - Wakayama Medical University Hospital, Wakayama
  - Yokohama City University Medical Center, Yokohama
- Jordan (4):
  - Khalidi Hospital and Medical Center, Amman
  - Jordan University Hospital, Amman
  - Irbid Specialty Hospital, Irbid
  - King Abdullah University Hospital, Irbid
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, Riga
  - Alda Pukisa arsta prakse, Riga
- Lebanon (8):
  - Ain Wazein Hospital, Ain Wazein
  - American Universitty of Beirut Medical Center, Beirut
  - St Georges Hospital university medical centre, Beirut
  - Hotel Dieu de France Hospital, Beirut
  - Bellevue Medical Center, Beirut
  - Mount Lebanon Hospital, Beirut
  - Rafik Hariri University Hospital, Beirut
  - Nini Hospital, Tripoli
- Lithuania (2):
  - Lietuvos sveikatos mokslų universiteto ligoninė Kauno klinik, Kaunas
  - Vilnius University Hospital Santaros Klinikos, Public Institution, Vilnius
- Malaysia (6):
  - Hospital Ampang, Ampang
  - Hospital Raja Permaisuri Bainun, Ipoh
  - Hospital Sultanah Aminah, Johor Bharu
  - Hospital Raja Perempuan Zainab Ii, Kota Bharu
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
- Netherlands (3):
  - Amsterdam UMC locatie VUMC, Amsterdam
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Stichting Zuyderland Medisch Centrum, Sittard-Geleen
- New Zealand (4):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
- North Macedonia (2):
  - General City Hospital 8mi Septemvri, Skopje
  - University Clinic of Gastroenterohepatology, Skopje
- Poland (45):
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - Centrum Medyczne Lukamed, Chojnice
  - Synexus Polska Sp. z o.o. Oddzial w Czestochowie, Częstochowa
  - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk
  - Synexus Scm Sp Z o o Oddzial Gdynia, Gdynia
  - Prywatna Praktyka Lekarska, Jelenia Góra
  - Synexus Polska Sp z o o Oddzial w Katowicach, Katowice
  - Malopolskie Centrum Kliniczne, Krakow
  - Centrum Medyczne Plejady, Krakow
  - Centrum Medyczne Promed, Krakow
  - Centrum Opieki Zdrowotnej Orkan Med Stec Michalska sj, Ksawerów
  - Synexus Polska Sp z o o, Lodz
  - AmiCare Centrum Medyczne, Lodz
  - 1 Wojskowy Szpital Kliniczny Z Poliklinika SPZOZ W Lublinie, Lublin
  - Gastromed Spotka Z Ograniczona Odpowiedzialnoscia Sp. K., Lublin
  - Wojewodzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - Twoja Przychodnia, Opole
  - Oswiecimskie Centrum Badan Klinicznych, Oświęcim
  - EMC Instytut Medyczny SA, Poznan
  - Solumed S C, Poznan
  - Synexus Polska Sp. z.o.o. Oddzial w Poznaniu, Poznan
  - Twoja Przychodnia, Poznan
  - Centrum Medyczne 'Medyk' Sp. z o.o. K., Rzeszów
  - Endoskopia Sp z o.o., Sopot
  - Kiepury Clinic, Sosnowiec
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - Niepubliczny Zaklad Opieki Zdrowotnej, Szczecin
  - GASTROMED Specjalistyczne Centrum Gastrologii i Endoskopii Specjalistyczne Gabinety Lekarskie, Torun
  - H-T Centrum Medyczne Endoterapia, Tychy
  - Wojskowy Instytut Medyczny, Warsaw
  - Centrum Medyczne, Warsaw
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw
  - Centrum Badawcze Wspolczesnej Terapii, Warsaw
  - NZOZ Vivamed Zespol Lekarzy Specjalistow, Warsaw
  - Szpital Pomnik Centrum Zdrowia Dziecka, Warsaw
  - Synexus Polska Sp z o o Oddzial w Warszawie, Warsaw
  - Centrum Zdrowia Tuchow, Wierzchosławice
  - Synexus Polska Sp z o o Oddzial we Wroclawiu, Wroclaw
  - Przychodnia Vistamed, Wroclaw
  - Futuremeds sp. z o.o., Wroclaw
  - Melita Medical Sp. z o.o., Wroclaw
  - ARS MEDICA Rybak Maria, Rybak Zbigniew, s.c., Wroclaw
  - EuroMediCare Szpital Specjalistyczny z Przychodnia, Wroclaw
  - Centrum Diagnostyczno - Lecznicze Barska sp. z o.o. Szpital Specjalistyczny Barska, Włocławek
  - ETG Zamosc, Zamość
- Portugal (6):
  - Hospital de Braga, Braga
  - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - Uls Alto Ave - Hosp. Sra. Da Oliveira Guimaraes, Guimarães
  - Hospital de Portimao-Centro Hospitalar do Barlavento Algarvio, Portimão
  - H. Santo António - Centro Hospitalar do Porto, Porto
  - Centro Hospitalar de Entre o Douro e Vouga, E.P.E, Santa Maria da Feira
- San Juan Bautista School of Medicine, Caguas, Puerto Rico
- Russia (21):
  - Kazan State Medical University, Kazan'
  - KGBUZ 'Regional Clinical Hospital', Krasnoyarsk
  - State Scientific Centre of Coloproctology, Moscow
  - Novgorod Regional Clinical Hospital n.a. N.A. Semashko, Nizhny Novgorod
  - City Clinical Hospital #12, Novosibirsk
  - FSBI 'Scientific Research Institute of Clinical and Experimental Lymphology' of Siberian Branch, Novosibirsk
  - Clinical Diagnostic Center 'Ultramed', Omsk
  - GBUZ of Moscow Region City Clinical Hospital #3, Podolsk
  - GBOU VPO Rostov State Medical University, Rostov-on-Don
  - City Hospital #20, Rostov-on-Don
  - Clinical Hospital #122 n.a. after L.G. Sokolov, Saint Petersburg
  - City Hospital named after St. Martyr Elizabeth, Saint Petersburg
  - The Limited Liability Company Research center Eco-safety, Saint Petersburg
  - St.Petersburg State Medical University n.a.Pavlov, Saint Petersburg
  - City Clinical Hospital #31, Saint Petersburg
  - Medical University Reaviz, Samara
  - NUZ 'Railway Clinical Hospital on Samara station of LLC 'Russian Railways', Samara
  - Saratov City Hospital #5, Saratov
  - Tomsk Regional Clinical Hospital, Tomsk
  - Ulyanovsk Regional Clinical Hospital, Ulyanovsk
  - GUZ Novgorod Regional Clinical Hospital, Veliky Novgorod
- Saudi Arabia (2):
  - King Abdullah Medical City in Holy Capital, Mecca
  - King Abdul Aziz Medical City for National Guard Health Affairs, Riyadh
- Serbia (6):
  - Special hospital for Internal diseases, Oncomed system, Belgrade
  - University Clinical Center of Serbia, Belgrade
  - Zvezdara University Medical Center, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
  - General Hospital 'Djordje Joanovic', Zrenjanin
- Slovakia (3):
  - FNsP F.D.R. Banska Bystrica, Banská Bystrica
  - ENDOMED s.r.o, Košice
  - GASTRO I. s.r.o., Prešov
- South Korea (18):
  - Korea University Ansan Hospital, Ansan-si
  - Inje University Haeundae Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Kyongpook national university Medical center, Daegu
  - Kyungpook National University Hospital, Daegu
  - The Catholic university of Korea, St. Vincent's Hospital, Gyeonggi-do
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si
  - CHA Bundang Medical Center, CHA University, Seongnam
  - The Catholic Univ of Korea DaeJeon St Mary s Hospital, Seongnam
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kangbuk Samsung Hospital, Seoul
  - Yonsei University College of Medicine, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Wonju Christian Hospital, Wŏnju
  - Ewha Womans University Mokdong Hospital, Yangch’ŏn-gu
- Spain (11):
  - Hosp Reina Sofia, Córdoba
  - Complejo Hosp Univ. de Ferrol, Ferrol
  - Hosp. Univ. Dr. Josep Trueta, Girona
  - Hosp. Gral. Juan Ramon Jimenez, Huelva
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Univ. Central de Asturias, Oviedo
  - Hosp. Provincial de Pontevedra, Pontevedra
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Univ. de Torrejon, Torrejón de Ardoz
  - Hosp. Alvaro Cunqueiro, Vigo
  - Hosp. Univ. Miguel Servet, Zaragoza
- Taiwan (4):
  - Chang-Hua Christian Hospital, Changhua
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang-Gung Memorial Hospital-Linkou, Taoyuan District
- Tunisia (5):
  - Hopital Regional Mohamed Tahar El Maamouri, Nabeul
  - Hopital Universitaire Sahloul, Sousse
  - Hopital Habib Thameur, Tunis
  - Military Hospital of Instruction of Tunis, Tunis
  - Hospital La Rabta, Tunis Jebbari
- Turkey (Türkiye) (9):
  - Hacettepe University Medical Faculty, Ankara
  - Gulhane Egitim ve Arastirma Hastanesi, Ankara
  - Firat University Hospital, Elâzığ
  - Mustafa Kemal University Research and Practise Hospital, Hatay
  - Acibadem Fulya Hospital, Istanbul
  - Sisli Etfal Egitim ve Arastirma Hospital, Istanbul
  - BAU Medical Park Goztepe Hospital, Istanbul
  - Marmara University Medical Faculty, Istanbul
  - Dokuz Eylul University Medical Faculty, Izmir
- Ukraine (13):
  - MNCE City Clinical Hospital No 2 named after prof O O Shalimov of the Kharkiv City Council, Kharkiv
  - SE 'National institute therapy named L.T. Maloi NAMS of Ukraine', Kharkiv
  - KZ Khersonska Miska Klinichna Likarnia Im. Ye.Ie.Karabelesha, Kherson
  - KNP Kyivska miska klinichna likarnia №18 vykonavchoho orhanu KMR (KMDA), Kyiv
  - LLC Treatment and Diagnostic Center Adonis Plus, Kyiv
  - Medical Research and Practice Center Medbud of the Public Joint Stock Holding Company Kyivmiskbud, Kyiv
  - Kyiv Railway Clinical Hospital #2 Of Branch 'Health Center' Of The Company 'Ukrainian Railway', Kyiv
  - Kyiv Regional Clinical Hospital, Kyiv
  - Odeska oblasna klinichna likarnia, Odesa
  - Ternopil municipal hospital #1, Ternopil
  - MNCE Zakarpatska Regional Clinical Hospital named after A Novak of Zakarpatska Regional Council, Uzhhorod
  - Health Clinic Limited Liability Company, Vinnytsia
  - KU 6 miska klinichna likarnia ZMR, Zaporizhzhya
- United Kingdom (3):
  - Barnsley District General Hospital, Barnsley
  - Addenbrooke's Hospital, Cambridge
  - St Georges Healthcare NHS Trust, London

REFERENCES:
- [Derived] Panaccione R, Feagan BG, Afzali A, Rubin DT, Reinisch W, Panes J, Danese S, Hisamatsu T, Terry NA, Salese L, Van Rampelbergh R, Sahoo A, Vetter ML, Yee J, Han C, Frustaci ME, Wan KYY, Yang Z, Johanns J, Andrews JM, D'Haens GR, Sands BE; GALAXI 2 & 3 Study Group. Efficacy and safety of intravenous induction and subcutaneous maintenance therapy with guselkumab for patients with Crohn's disease (GALAXI-2 and GALAXI-3): 48-week results from two phase 3, randomised, placebo and active comparator-controlled, double-blind, triple-dummy trials. Lancet. 2025 Jul 26;406(10501):358-375. doi: 10.1016/S0140-6736(25)00681-6. Epub 2025 Jul 17. PMID 40684778
- [Derived] Hasskamp J, Meinhardt C, Timmer A. Anti-IL-12/23p40 antibodies for induction of remission in Crohn's disease. Cochrane Database Syst Rev. 2025 May 13;5(5):CD007572. doi: 10.1002/14651858.CD007572.pub4. PMID 40357993
- [Derived] Danese S, Panaccione R, Feagan BG, Afzali A, Rubin DT, Sands BE, Reinisch W, Panes J, Sahoo A, Terry NA, Chan D, Han C, Frustaci ME, Yang Z, Sandborn WJ, Hisamatsu T, Andrews JM, D'Haens GR; GALAXI-1 Study Group. Efficacy and safety of 48 weeks of guselkumab for patients with Crohn's disease: maintenance results from the phase 2, randomised, double-blind GALAXI-1 trial. Lancet Gastroenterol Hepatol. 2024 Feb;9(2):133-146. doi: 10.1016/S2468-1253(23)00318-7. Epub 2023 Dec 14. PMID 38104569
- [Derived] Sandborn WJ, D'Haens GR, Reinisch W, Panes J, Chan D, Gonzalez S, Weisel K, Germinaro M, Frustaci ME, Yang Z, Adedokun OJ, Han C, Panaccione R, Hisamatsu T, Danese S, Rubin DT, Sands BE, Afzali A, Andrews JM, Feagan BG; GALAXI-1 Investigators. Guselkumab for the Treatment of Crohn's Disease: Induction Results From the Phase 2 GALAXI-1 Study. Gastroenterology. 2022 May;162(6):1650-1664.e8. doi: 10.1053/j.gastro.2022.01.047. Epub 2022 Feb 5. PMID 35134323

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of 3 separate studies: Phase 2 dose-ranging study (GALAXI 1) and 2 identical Phase 3 confirmatory studies (GALAXI 2 and GALAXI 3). Participants with moderately to severely active Crohn's disease were enrolled in these studies.
Pre-assignment Details: Results were presented through Week 48 with a data cutoff date of 20 August 2020 (GALAXI 1), 20 October 2023 (GALAXI 2) and 16 October 2023 (GALAXI 3). At Week 48, participants who continued to benefit from treatment entered long-term extension period and continued to receive maintenance dose up to Week 236 which is still ongoing. Results of remaining duration of the study will be reported after study completion.
Groups:
- GALAXI 1 (Group 1) Guselkumab 1200 mg IV q4w Followed by 200 mg SC q4w: Participants received guselkumab 1200 milligrams (mg) intravenous (IV) infusion as induction dose at Weeks 0, 4 and 8. Participants then received guselkumab 200 mg subcutaneous (SC) injection every 4 weeks (q4w) as maintenance dose from Week 12 through Week 44.
- GALAXI 1 (Group 2) Guselkumab 600 mg IV q4w Followed by 200 mg SC q4w: Participants received guselkumab 600 mg IV infusion as induction dose at Weeks 0, 4 and 8. Participants then received guselkumab 200 mg SC injection q4w as maintenance dose from Week 12 through Week 44.
- GALAXI 1 (Group 3) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w: Participants received guselkumab 200 mg IV infusion as induction dose at Weeks 0, 4 and 8. Participants then received guselkumab 100 mg SC injection every 8 weeks (q8w) as maintenance dose from Week 16 through Week 40.
- GALAXI 1 (Group 4) Ustekinumab 6 mg/kg IV Followed by 90 mg SC q8w: Participants received a single weight-based dose of ustekinumab 6 milligrams per kilogram (mg/kg) IV infusion as induction dose at Week 0. From Week 8, participants received ustekinumab 90 mg SC injection q8w as maintenance dose through Week 40.
- GALAXI 1 (Group 5) Placebo q4w Followed by Placebo q4w or Ustekinumab 6mg/kg IV Then 90mg SC q8w: Participants received placebo (matching to guselkumab) IV infusion at Weeks 0, 4 and 8. At Week 12, participants were evaluated for clinical response (CR) (decrease from baseline in Crohn's Disease Activity Index [CDAI] score of greater than or equal to [>=] 100 points or CDAI score less than [<] 150). Participants who achieved CR at Week 12 continued to receive placebo q4w from Week 12 through Week 44. Participants who did not achieve CR at Week 12 received weight-based dose of ustekinumab 6 mg/kg IV infusion as induction dose at Week 12 followed by 90 mg SC injection q8w as maintenance dose from Week 20 through Week 44.
- GALAXI 2 (Group 1) Guselkumab 200 mg IV q4w Followed by 200 mg SC q4w; GALAXI 3 (Group 1) Guselkumab 200 mg IV q4w Followed by 200 mg SC q4w: Participants received guselkumab 200 mg IV infusion as induction dose at Weeks 0, 4 and 8. Participants then received guselkumab 200 mg SC injection q4w as maintenance dose from Week 12 through Week 44.
- GALAXI 2 (Group 2) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w; GALAXI 3 (Group 2) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w: Participants received guselkumab 200 mg IV infusion as induction dose at Weeks 0, 4 and 8. Participants then received guselkumab 100 mg SC injection q8w as maintenance dose from Week 16 through Week 40.
- GALAXI 2 (Group 3) Ustekinumab 6 mg/kg IV Followed by 90 mg SC q8w; GALAXI 3 (Group 3) Ustekinumab 6 mg/kg IV Followed by 90 mg SC q8w: Participants received a single weight-based dose of ustekinumab 6 mg/kg IV infusion as induction dose at Week 0. From Week 8, participants received ustekinumab 90 mg SC injection q8w as maintenance dose through Week 40.
- GALAXI 2 (Group 4) Placebo q4w Followed by Placebo q4w or Ustekinumab 6 mg/kg IV Then 90 mg SC q8w; GALAXI 3 (Group 4) Placebo q4w Followed by Placebo q4w or Ustekinumab 6 mg/kg IV Then 90 mg SC q8w: Participants received placebo (matching to guselkumab) IV infusion at Weeks 0, 4 and 8. At Week 12, participants were evaluated for CR (decrease from baseline in CDAI score of >=100 points or CDAI score <150). Participants who achieved CR at Week 12 continued to receive placebo q4w from Week 12 through Week 44. Participants who did not achieve CR at Week 12 received weight-based dose of ustekinumab 6 mg/kg IV infusion as induction dose at Week 12 followed by 90 mg SC injection q8w as maintenance dose from Week 20 through Week 44.
Period: Overall Study
Arm/Group | GALAXI 1 (Group 1) Guselkumab 1200 mg IV q4w Followed by 200 mg SC q4w | GALAXI 1 (Group 2) Guselkumab 600 mg IV q4w Followed by 200 mg SC q4w | GALAXI 1 (Group 3) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w | GALAXI 1 (Group 4) Ustekinumab 6 mg/kg IV Followed by 90 mg SC q8w | GALAXI 1 (Group 5) Placebo q4w Followed by Placebo q4w or Ustekinumab 6mg/kg IV Then 90mg SC q8w | GALAXI 2 (Group 1) Guselkumab 200 mg IV q4w Followed by 200 mg SC q4w | GALAXI 2 (Group 2) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w | GALAXI 2 (Group 3) Ustekinumab 6 mg/kg IV Followed by 90 mg SC q8w | GALAXI 2 (Group 4) Placebo q4w Followed by Placebo q4w or Ustekinumab 6 mg/kg IV Then 90 mg SC q8w | GALAXI 3 (Group 1) Guselkumab 200 mg IV q4w Followed by 200 mg SC q4w | GALAXI 3 (Group 2) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w | GALAXI 3 (Group 3) Ustekinumab 6 mg/kg IV Followed by 90 mg SC q8w | GALAXI 3 (Group 4) Placebo q4w Followed by Placebo q4w or Ustekinumab 6 mg/kg IV Then 90 mg SC q8w
Started | 73 | 73 | 73 | 71 | 70 | 148 | 149 | 150 | 77 | 151 | 148 | 150 | 76
Participants Who Did Not Achieve CR at Week 12 and Crossed Over to Ustekinumab | 0 | 0 | 0 | 0 | 43 | 0 | 0 | 0 | 49 | 0 | 0 | 0 | 51
Completed | 58 | 64 | 64 | 66 | 62 | 145 | 141 | 140 | 71 | 138 | 131 | 137 | 69
Not Completed | 15 | 9 | 9 | 5 | 8 | 3 | 8 | 10 | 6 | 13 | 17 | 13 | 7
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 14 | 7 | 8 | 4 | 6 | 3 | 6 | 9 | 6 | 11 | 14 | 12 | 7
Not completed — Other | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Randomized but not Treated | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics data were presented for all randomized participants who received at least 1 dose of study intervention.
Groups:
- GALAXI 1 (Group 1) Guselkumab 1200 mg IV q4w Followed by 200 mg SC q4w: Participants received guselkumab 1200 mg IV infusion as induction dose at Weeks 0, 4 and 8. Participants then received guselkumab 200 mg SC injection q4w as maintenance dose from Week 12 through Week 44.
- GALAXI 1 (Group 3) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w; GALAXI 2 (Group 2) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w; GALAXI 3 (Group 2) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w: Participants received guselkumab 200 mg IV infusion as induction dose at Weeks 0, 4 and 8. Participants then received guselkumab 100 mg SC injection q8w as maintenance dose from Week 16 through Week 40.
- GALAXI 1 (Group 4) Ustekinumab 6 mg/kg IV Followed by 90 mg SC q8w; GALAXI 2 (Group 3) Ustekinumab 6 mg/kg IV Followed by 90 mg SC q8w; GALAXI 3 (Group 3) Ustekinumab 6 mg/kg IV Followed by 90 mg SC q8w: Participants received a single weight-based dose of ustekinumab 6 mg/kg IV infusion as induction dose at Week 0. From Week 8, participants received ustekinumab 90 mg SC injection q8w as maintenance dose through Week 40.
- GALAXI 1 (Group 5) Placebo q4w Followed by Placebo q4w or Ustekinumab 6mg/kg IV Then 90mg SC q8w; GALAXI 2 (Group 4) Placebo q4w Followed by Placebo q4w or Ustekinumab 6 mg/kg IV Then 90 mg SC q8w; GALAXI 3 (Group 4) Placebo q4w Followed by Placebo q4w or Ustekinumab 6 mg/kg IV Then 90 mg SC q8w: Participants received placebo (matching to guselkumab) IV infusion at Weeks 0, 4 and 8. At Week 12, participants were evaluated for CR (decrease from baseline in CDAI score of >=100 points or CDAI score <150). Participants who achieved CR at Week 12 continued to receive placebo q4w from Week 12 through Week 44. Participants who did not achieve CR at Week 12 received weight-based dose of ustekinumab 6 mg/kg IV infusion as induction dose at Week 12 followed by 90 mg SC injection q8w as maintenance dose from Week 20 through Week 44.
- Total: Total of all reporting groups
Arm/Group | GALAXI 1 (Group 1) Guselkumab 1200 mg IV q4w Followed by 200 mg SC q4w | GALAXI 1 (Group 2) Guselkumab 600 mg IV q4w Followed by 200 mg SC q4w | GALAXI 1 (Group 3) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w | GALAXI 1 (Group 4) Ustekinumab 6 mg/kg IV Followed by 90 mg SC q8w | GALAXI 1 (Group 5) Placebo q4w Followed by Placebo q4w or Ustekinumab 6mg/kg IV Then 90mg SC q8w | GALAXI 2 (Group 1) Guselkumab 200 mg IV q4w Followed by 200 mg SC q4w | GALAXI 2 (Group 2) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w | GALAXI 2 (Group 3) Ustekinumab 6 mg/kg IV Followed by 90 mg SC q8w | GALAXI 2 (Group 4) Placebo q4w Followed by Placebo q4w or Ustekinumab 6 mg/kg IV Then 90 mg SC q8w | GALAXI 3 (Group 1) Guselkumab 200 mg IV q4w Followed by 200 mg SC q4w | GALAXI 3 (Group 2) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w | GALAXI 3 (Group 3) Ustekinumab 6 mg/kg IV Followed by 90 mg SC q8w | GALAXI 3 (Group 4) Placebo q4w Followed by Placebo q4w or Ustekinumab 6 mg/kg IV Then 90 mg SC q8w | Total
Number analyzed (Participants) | 73 | 73 | 73 | 71 | 70 | 148 | 148 | 150 | 77 | 151 | 148 | 150 | 76 | 1408
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 68 | 66 | 69 | 69 | 68 | 142 | 144 | 143 | 76 | 143 | 146 | 143 | 75 | 1352
  >=65 years | 5 | 7 | 4 | 2 | 2 | 6 | 4 | 7 | 1 | 8 | 2 | 7 | 1 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.2 (14.28) | 39.3 (15.51) | 41.5 (14.41) | 36.3 (12.08) | 39 (12.79) | 36.2 (13.03) | 37.3 (12.86) | 37 (12.76) | 34.1 (11.81) | 37.6 (13.4) | 34.8 (11.48) | 37.9 (13.61) | 35.8 (12.48) | 37.2 (13.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 29 | 27 | 26 | 26 | 59 | 76 | 62 | 35 | 59 | 60 | 66 | 26 | 586
  Male | 38 | 44 | 46 | 45 | 44 | 89 | 72 | 88 | 42 | 92 | 88 | 84 | 50 | 822
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 4 | 0 | 4 | 8 | 5 | 7 | 2 | 5 | 7 | 11 | 4 | 65
  Not Hispanic or Latino | 69 | 64 | 66 | 69 | 64 | 136 | 139 | 137 | 71 | 142 | 136 | 131 | 71 | 1295
  Unknown or Not Reported | 1 | 4 | 3 | 2 | 2 | 4 | 4 | 6 | 4 | 4 | 5 | 8 | 1 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Asian | 6 | 10 | 9 | 8 | 5 | 28 | 34 | 32 | 17 | 28 | 38 | 23 | 19 | 257
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 11
  Black or African American | 2 | 2 | 0 | 1 | 3 | 1 | 3 | 3 | 0 | 1 | 0 | 4 | 3 | 23
  White | 61 | 59 | 58 | 61 | 58 | 117 | 108 | 111 | 56 | 118 | 107 | 116 | 50 | 1080
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3 | 0 | 4 | 2 | 3 | 4 | 2 | 4 | 2 | 6 | 2 | 35
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 1 | 0 | 0 | 0 | 0 | 5 | 2 | 6 | 1 | 2 | 1 | 3 | 1 | 22
  Austria | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Belarus | 2 | 1 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 10
  Belgium | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 5
  Bosnia and Herzegovina | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 3 | 1 | 0 | 2 | 2 | 0 | 14
  Brazil | 0 | 0 | 0 | 0 | 0 | 6 | 7 | 9 | 2 | 8 | 6 | 12 | 3 | 53
  Canada | 0 | 0 | 2 | 0 | 0 | 1 | 6 | 4 | 1 | 2 | 4 | 5 | 2 | 27
  China | 0 | 0 | 0 | 0 | 0 | 18 | 19 | 10 | 12 | 15 | 22 | 12 | 12 | 120
  Colombia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Croatia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 4
  Czech Republic | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 3 | 1 | 4 | 1 | 1 | 16
  France | 2 | 2 | 6 | 1 | 2 | 4 | 2 | 4 | 2 | 1 | 1 | 2 | 1 | 30
  Georgia | 1 | 3 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 10
  Germany | 3 | 4 | 0 | 2 | 2 | 2 | 4 | 2 | 0 | 4 | 2 | 1 | 1 | 27
  Greece | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hungary | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 5 | 0 | 4 | 1 | 4 | 1 | 20
  India | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 2 | 2 | 0 | 10
  Israel | 2 | 2 | 2 | 2 | 0 | 4 | 1 | 0 | 2 | 0 | 9 | 0 | 2 | 26
  Italy | 2 | 2 | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 3 | 1 | 0 | 1 | 15
  Japan | 3 | 5 | 6 | 4 | 2 | 4 | 7 | 13 | 1 | 9 | 6 | 4 | 4 | 68
  Jordan | 1 | 1 | 0 | 2 | 1 | 4 | 3 | 4 | 4 | 9 | 3 | 9 | 1 | 42
  Latvia | 3 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 10
  Lebanon | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 1 | 1 | 2 | 3 | 4 | 2 | 19
  Lithuania | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Malaysia | 1 | 2 | 0 | 1 | 0 | 3 | 1 | 2 | 1 | 0 | 2 | 1 | 1 | 15
  Netherlands | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 4 | 1 | 2 | 0 | 12
  New Zealand | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 3 | 1 | 2 | 1 | 0 | 0 | 12
  Poland | 11 | 18 | 15 | 21 | 25 | 33 | 24 | 33 | 10 | 26 | 32 | 28 | 16 | 292
  Portugal | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 4
  Macedonia | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 9
  Russian Federation | 6 | 3 | 8 | 4 | 3 | 14 | 14 | 14 | 10 | 13 | 9 | 9 | 8 | 115
  Saudi Arabia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Slovakia | 1 | 1 | 0 | 2 | 2 | 1 | 3 | 1 | 0 | 3 | 2 | 1 | 0 | 17
  Korea, South | 1 | 2 | 1 | 3 | 2 | 2 | 5 | 4 | 2 | 2 | 3 | 3 | 2 | 32
  Spain | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 3 | 0 | 12
  Serbia | 2 | 3 | 3 | 6 | 2 | 8 | 9 | 7 | 3 | 5 | 2 | 8 | 6 | 64
  Taiwan | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 7
  Tunisia | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 1 | 1 | 5 | 2 | 1 | 1 | 19
  Turkey | 1 | 1 | 0 | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 10
  Ukraine | 9 | 7 | 7 | 7 | 6 | 11 | 12 | 7 | 8 | 11 | 10 | 7 | 4 | 106
  United Kingdom | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 5
  United States | 14 | 10 | 13 | 6 | 14 | 7 | 6 | 8 | 2 | 10 | 9 | 15 | 5 | 119

OUTCOME MEASURES:

1. Primary Outcome: GALAXI 1: Change From Baseline in the Crohn's Disease Activity Index (CDAI) Score at Week 12
Description: The multi-item CDAI score assessed severity of illness by collecting information on 8 different Crohn's disease-related variables (extraintestinal manifestations, abdominal mass, weight, hematocrit, use of antidiarrheal drug(s) and/or opiates, total number of liquid or very soft stools, abdominal pain/cramps, and general well-being). The last 3 variables were scored over 7 eligible days by the participant on a diary card. The total CDAI score ranged from 0 to 600 in general: higher score indicated higher disease activities. A decrease in total CDAI score over time indicates improvement in disease activity. Baseline was defined as the last observation prior to or at the date of the first study intervention.
Time Frame: Baseline and Week 12
Population: The primary efficacy analysis set consisted of randomized participants who received at least 1 dose of study intervention (including a partial dose), except for those participants whose induction dosing was discontinued as a result of the urgent safety measure. Here 'N' (overall number of participants analyzed) refers to the number of participants evaluable for this outcome measure. This outcome measure was planned to be collected and analyzed for specified arms only.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- GALAXI 1 (Group 5) Placebo q4w Followed by Placebo q4w: Participants received placebo (matching to guselkumab) IV infusion at Weeks 0, 4 and 8. At Week 12, participants were evaluated for CR (decrease from baseline in CDAI score of >=100 points or CDAI score <150). Participants who achieved CR at Week 12 continued to receive placebo q4w from Week 12 through Week 44.
Arm/Group | GALAXI 1 (Group 1) Guselkumab 1200 mg IV q4w Followed by 200 mg SC q4w | GALAXI 1 (Group 2) Guselkumab 600 mg IV q4w Followed by 200 mg SC q4w | GALAXI 1 (Group 3) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w | GALAXI 1 (Group 5) Placebo q4w Followed by Placebo q4w
Number analyzed (Participants) | 58 | 62 | 60 | 60
Units on a scale | -143.7 (96.58) | -139.2 (100.71) | -159.8 (110.52) | -34.4 (104.85)
Statistical Analysis 1: Comparison: GALAXI 1 (Group 3) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w vs GALAXI 1 (Group 5) Placebo q4w Followed by Placebo q4w; Test type: Superiority; p < 0.001, Mixed Model for Repeated Measure; Least Square (LS) Mean Difference = 124.2, 95% CI 2-sided [89.8 to 158.7] — LS Mean difference between the treatment groups and p-values for the comparisons of each guselkumab treatment group with the placebo group were based on MMRM analysis
Statistical Analysis 2: Comparison: GALAXI 1 (Group 2) Guselkumab 600 mg IV q4w Followed by 200 mg SC q4w vs GALAXI 1 (Group 5) Placebo q4w Followed by Placebo q4w; Test type: Superiority; p < 0.001, Mixed Model for Repeated Measure; LS Mean Difference = 102.7, 95% CI 2-sided [68.5 to 136.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: GALAXI 1 (Group 1) Guselkumab 1200 mg IV q4w Followed by 200 mg SC q4w vs GALAXI 1 (Group 5) Placebo q4w Followed by Placebo q4w; Test type: Superiority; p < 0.001, Mixed Model for Repeated Measure; LS Mean Difference = 108.7, 95% CI 2-sided [73.9 to 143.5] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Global: GALAXI 2: Percentage of Participants With Both Clinical Response at Week 12 and Clinical Remission at Week 48
Description: Clinical response was defined as a decrease from baseline (BL) in CDAI score greater than or equal to (>=) 100 points or CDAI score <150. Clinical remission was defined as a CDAI score <150. The multi-item CDAI score assessed severity of illness by collecting information on 8 different Crohn's disease-related variables (extraintestinal manifestations, abdominal mass, weight, hematocrit, use of antidiarrheal drug(s) and/or opiates, total number of liquid or very soft stools, abdominal pain/cramps, and general well-being). The last 3 variables were scored over 7 eligible days by the participant on a diary card. The total CDAI score ranged from 0 to 600 in general: higher score indicated higher disease activities. A decrease in total CDAI score over time indicates improvement in disease activity.
Time Frame: Weeks 48
Population: The primary analysis set included all randomized participants who received at least 1 (partial or complete) dose of study intervention and satisfied the simple endoscopic score for crohn's disease (SES-CD) eligibility criteria (that is, screening SES-CD score >=6 [or >=4 for participants with isolated ileal disease]). Data were planned to be collected and analyzed for specified arms only.
Measure: Number; unit: Percentage of participants
Arm/Group | GALAXI 2 (Group 1) Guselkumab 200 mg IV q4w Followed by 200 mg SC q4w | GALAXI 2 (Group 2) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w | GALAXI 2 (Group 4) Placebo q4w Followed by Placebo q4w or Ustekinumab 6 mg/kg IV Then 90 mg SC q8w
Number analyzed (Participants) | 146 | 143 | 76
Percentage of participants | 54.8 | 49.0 | 11.8
Statistical Analysis 1: Comparison: GALAXI 2 (Group 2) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w vs GALAXI 2 (Group 4) Placebo q4w Followed by Placebo q4w or Ustekinumab 6 mg/kg IV Then 90 mg SC q8w; Test type: Superiority; p < 0.001, Mantel Haenszel; Adjusted treatment difference = 38.1, 95% CI 2-sided [27.3 to 48.9] — Treatment difference between guselkumab group and placebo group was based on the common risk difference by use of Mantel- Haenszel stratum weights and the Sato variance estimator
Statistical Analysis 2: Comparison: GALAXI 2 (Group 1) Guselkumab 200 mg IV q4w Followed by 200 mg SC q4w vs GALAXI 2 (Group 4) Placebo q4w Followed by Placebo q4w or Ustekinumab 6 mg/kg IV Then 90 mg SC q8w; Test type: Superiority; p < 0.001, Mantel Haenszel; Adjusted treatment difference = 42.8, 95% CI 2-sided [31.6 to 53.9] — Treatment difference between guselkumab group and placebo group was based on the common risk difference by use of Mantel-Haenszel stratum weights and the Sato variance estimator

3. Primary Outcome: Global: GALAXI 2: Percentage of Participants With Both Clinical Response (CR) at Week 12 and Endoscopic Response (ER) at Week 48
Description: CR: decrease from BL in CDAI score >=100/<150. ER: >=50% improvement from BL in SES-CD score/SES-CD score <=2. CDAI(8 variables):extraintestinal manifestations, abdominal mass, weight, hematocrit, use of antidiarrheal drug(s) and/or opiates, total number of liquid/soft stools, abdominal pain/cramps, general well-being. Last 3 variables scored over 7 eligible days by participant on diary. Total CDAI score ranged:0-600(in general):higher score=higher disease activities. Decrease in total CDAI score over time=improvement in disease. SES-CD evaluated 4 endoscopic components (presence & size of ulcer, extent of ulcerated surface, extent of affected surface, presence & type of narrowing) across 5 ileocolonic segments (ileum; right, left & transverse colon; rectum) each scored 0(best) to 3(worst) except narrowing component for which maximum total score (that is, stricturing) was 11 points. SES-CD score: sum of all component scores(all segments) ranged:0-56, higher scores=more severe disease.
Time Frame: Weeks 48
Population: The primary analysis set included all randomized participants who received at least 1 (partial or complete) dose of study intervention and satisfied the SES-CD eligibility criteria (that is, screening SES-CD score >=6 [or >=4 for participants with isolated ileal disease]). Data were planned to be collected and analyzed for specified arms only.
Measure: Number; unit: Percentage of participants
Arm/Group | GALAXI 2 (Group 1) Guselkumab 200 mg IV q4w Followed by 200 mg SC q4w | GALAXI 2 (Group 2) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w | GALAXI 2 (Group 4) Placebo q4w Followed by Placebo q4w or Ustekinumab 6 mg/kg IV Then 90 mg SC q8w
Number analyzed (Participants) | 146 | 143 | 76
Percentage of participants | 38.4 | 39.2 | 5.3
Statistical Analysis 1: Comparison: GALAXI 2 (Group 2) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w vs GALAXI 2 (Group 4) Placebo q4w Followed by Placebo q4w or Ustekinumab 6 mg/kg IV Then 90 mg SC q8w; Test type: Superiority; p < 0.001, Mantel Haenszel; Adjusted treatment difference = 33.7, 95% CI 2-sided [24.1 to 43.2] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: GALAXI 2 (Group 1) Guselkumab 200 mg IV q4w Followed by 200 mg SC q4w vs GALAXI 2 (Group 4) Placebo q4w Followed by Placebo q4w or Ustekinumab 6 mg/kg IV Then 90 mg SC q8w; Test type: Superiority; p < 0.001, Mantel Haenszel; Adjusted treatment difference = 32.9, 95% CI 2-sided [23.5 to 42.4] — [estimate comment as in outcome 2, analysis 2]

4. Primary Outcome: Global: GALAXI 3: Percentage of Participants With Both Clinical Response at Week 12 and Clinical Remission at Week 48
Description: Clinical response was defined as a decrease from baseline in CDAI score >= 100 points or CDAI score <150. Clinical remission was defined as a CDAI score <150. The multi-item CDAI score assessed severity of illness by collecting information on 8 different Crohn's disease-related variables (extraintestinal manifestations, abdominal mass, weight, hematocrit, use of antidiarrheal drug(s) and/or opiates, total number of liquid or very soft stools, abdominal pain/cramps, and general well-being). The last 3 variables were scored over 7 eligible days by the participant on a diary card. The total CDAI score ranged from 0 to 600 in general: higher score indicated higher disease activities. A decrease in total CDAI score over time indicates improvement in disease activity.
Time Frame: Weeks 48
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | GALAXI 3 (Group 1) Guselkumab 200 mg IV q4w Followed by 200 mg SC q4w | GALAXI 3 (Group 2) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w | GALAXI 3 (Group 4) Placebo q4w Followed by Placebo q4w or Ustekinumab 6 mg/kg IV Then 90 mg SC q8w
Number analyzed (Participants) | 150 | 143 | 72
Percentage of participants | 48.0 | 46.9 | 12.5
Statistical Analysis 1: Comparison: GALAXI 3 (Group 2) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w vs GALAXI 3 (Group 4) Placebo q4w Followed by Placebo q4w or Ustekinumab 6 mg/kg IV Then 90 mg SC q8w; Test type: Superiority; p < 0.001, Mantel Haenszel; Adjusted treatment difference = 34.2, 95% CI 2-sided [23.2 to 45.3] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: GALAXI 3 (Group 1) Guselkumab 200 mg IV q4w Followed by 200 mg SC q4w vs GALAXI 3 (Group 4) Placebo q4w Followed by Placebo q4w or Ustekinumab 6 mg/kg IV Then 90 mg SC q8w; Test type: Superiority; p < 0.001, Mantel Haenszel; Adjusted treatment difference = 35, 95% CI 2-sided [23.5 to 46.5] — [estimate comment as in outcome 2, analysis 2]

5. Primary Outcome: Global: GALAXI 3: Percentage of Participants With Both Clinical Response (CR) at Week 12 and Endoscopic Response (ER) at Week 48
Description: as for outcome 3
Time Frame: Weeks 48
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | GALAXI 3 (Group 1) Guselkumab 200 mg IV q4w Followed by 200 mg SC q4w | GALAXI 3 (Group 2) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w | GALAXI 3 (Group 4) Placebo q4w Followed by Placebo q4w or Ustekinumab 6 mg/kg IV Then 90 mg SC q8w
Number analyzed (Participants) | 150 | 143 | 72
Percentage of participants | 36.0 | 33.6 | 5.6
Statistical Analysis 1: Comparison: GALAXI 3 (Group 2) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w vs GALAXI 3 (Group 4) Placebo q4w Followed by Placebo q4w or Ustekinumab 6 mg/kg IV Then 90 mg SC q8w; Test type: Superiority; p < 0.001, Mantel Haenszel; Adjusted treatment difference = 27.9, 95% CI 2-sided [18.7 to 37.1] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 2: Comparison: GALAXI 3 (Group 1) Guselkumab 200 mg IV q4w Followed by 200 mg SC q4w vs GALAXI 3 (Group 4) Placebo q4w Followed by Placebo q4w or Ustekinumab 6 mg/kg IV Then 90 mg SC q8w; Test type: Superiority; p < 0.001, Mantel Haenszel; Adjusted treatment difference = 30.8, 95% CI 2-sided [21.3 to 40.3] — [estimate comment as in outcome 2, analysis 2]

6. Primary Outcome: Regional: GALAXI 2: Percentage of Participants With Clinical Remission at Week 12
Description: Clinical remission was defined as a CDAI score <150. The multi-item CDAI score assessed severity of illness by collecting information on 8 different Crohn's disease-related variables (extraintestinal manifestations, abdominal mass, weight, hematocrit, use of antidiarrheal drug(s) and/or opiates, total number of liquid or very soft stools, abdominal pain/cramps, and general well-being). The last 3 variables were scored over 7 eligible days by the participant on a diary card. The total CDAI score ranged from 0 to 600 in general: higher score indicated higher disease activities. A decrease in total CDAI score over time indicates improvement in disease activity.
Time Frame: Week 12
Population: Primary analysis set: all randomized participants who received at least 1 (partial or complete) dose of study intervention and satisfied the SES-CD eligibility criteria (that is, screening SES-CD score >=6 [or >=4 for participants with isolated ileal disease]). Data for this outcome measure was planned to be collected and analyzed as a combined group for participants who received guselkumab induction dose in GALAXI 2 Groups 1 and 2, and for participants who received placebo in GALAXI 2 Group 4.
Measure: Number; unit: Percentage of participants
Groups:
- GALAXI 2 Placebo (From Group 4): Participants received placebo (matching to guselkumab) IV infusion at Weeks 0, 4 and 8.
- GALAXI 2 Combined Guselkumab 200 mg IV (Group 1+ Group 2): Participants received guselkumab 200 mg IV infusion at Weeks 0, 4, and 8.
Arm/Group | GALAXI 2 Placebo (From Group 4) | GALAXI 2 Combined Guselkumab 200 mg IV (Group 1+ Group 2)
Number analyzed (Participants) | 76 | 289
Percentage of participants | 22.4 | 47.1
Statistical Analysis 1: Comparison: GALAXI 2 Placebo (From Group 4) vs GALAXI 2 Combined Guselkumab 200 mg IV (Group 1+ Group 2); Test type: Superiority; p < 0.001, Mantel Haenszel; Adjusted treatment difference = 25.1, 95% CI 2-sided [14.1 to 36.2] — Treatment difference between combined guselkumab group and placebo group was based on the common risk difference by use of Mantel- Haenszel stratum weights and the Sato variance estimator

7. Primary Outcome: Regional: GALAXI 2: Percentage of Participants With Endoscopic Response at Week 12
Description: Endoscopic response was defined as >=50% improvement from baseline in SES-CD score or SES-CD score <=2. SES-CD evaluated 4 endoscopic components (presence and size of ulcer, extent of ulcerated surface, extent of affected surface, presence and type of narrowing) across 5 ileocolonic segments (ileum, right colon, transverse colon, left colon, rectum), each scored 0 (best) to 3 (worst) except narrowing component for which maximum total score (that is, stricturing) was 11 points. Total SES-CD score: sum of all component scores across all segments, ranged: 0 to 56, higher scores = more severe disease.
Time Frame: Week 12
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | GALAXI 2 Placebo (From Group 4) | GALAXI 2 Combined Guselkumab 200 mg IV (Group 1+ Group 2)
Number analyzed (Participants) | 76 | 289
Percentage of participants | 10.5 | 37.7
Statistical Analysis 1: Comparison: GALAXI 2 Placebo (From Group 4) vs GALAXI 2 Combined Guselkumab 200 mg IV (Group 1+ Group 2); Test type: Superiority; p < 0.001, Mantel Haenszel; Adjusted treatment difference = 27.7, 95% CI 2-sided [19.3 to 36.1] — [estimate comment as in outcome 6, analysis 1]

8. Primary Outcome: Regional: GALAXI 3: Percentage of Participants With Clinical Remission at Week 12
Description: as for outcome 6
Time Frame: Week 12
Population: Primary analysis set: all randomized participants who received at least 1 (partial or complete) dose of study intervention and satisfied the SES-CD eligibility criteria (that is, screening SES-CD score >=6 [or >=4 for participants with isolated ileal disease]). Data for this outcome measure was planned to be collected and analyzed as a combined group for participants who received guselkumab induction dose in GALAXI 3 Groups 1 and 2, and for participants who received placebo in GALAXI 3 Group 4.
Measure: Number; unit: Percentage of participants
Groups:
- GALAXI 3 Placebo (From Group 4): Participants received placebo (matching to guselkumab) IV infusion at Weeks 0, 4 and 8.
- GALAXI 3 Combined Guselkumab 200 mg IV (Group 1+ Group 2): Participants received guselkumab 200 mg IV infusion at Weeks 0, 4, and 8.
Arm/Group | GALAXI 3 Placebo (From Group 4) | GALAXI 3 Combined Guselkumab 200 mg IV (Group 1+ Group 2)
Number analyzed (Participants) | 72 | 293
Percentage of participants | 15.3 | 47.1
Statistical Analysis 1: Comparison: GALAXI 3 Placebo (From Group 4) vs GALAXI 3 Combined Guselkumab 200 mg IV (Group 1+ Group 2); Test type: Superiority; p < 0.001, Mantel Haenszel; Adjusted treatment difference = 31.2, 95% CI 2-sided [21.1 to 41.3] — [estimate comment as in outcome 6, analysis 1]

9. Primary Outcome: Regional: GALAXI 3: Percentage of Participants With Endoscopic Response at Week 12
Description: as for outcome 7
Time Frame: Week 12
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | GALAXI 3 Placebo (From Group 4) | GALAXI 3 Combined Guselkumab 200 mg IV (Group 1+ Group 2)
Number analyzed (Participants) | 72 | 293
Percentage of participants | 13.9 | 36.2
Statistical Analysis 1: Comparison: GALAXI 3 Placebo (From Group 4) vs GALAXI 3 Combined Guselkumab 200 mg IV (Group 1+ Group 2); Test type: Superiority; p < 0.001, Mantel Haenszel; Adjusted treatment difference = 22.1, 95% CI 2-sided [12.2 to 31.9] — [estimate comment as in outcome 6, analysis 1]

10. Secondary Outcome: GALAXI 1: Percentage of Participants With Clinical Remission at Week 12
Time Frame: At Week 12
Reporting Status: Not Posted, anticipated posting 2031-06

11. Secondary Outcome: GALAXI 1: Percentage of Participants With Clinical Response at Week 12
Time Frame: At Week 12
Reporting Status: Not Posted, anticipated posting 2031-06

12. Secondary Outcome: GALAXI 1: Percentage of Participants With Patient-Reported Outcome (PRO) 2 Remission at Week 12
Time Frame: At Week 12
Reporting Status: Not Posted, anticipated posting 2031-06

13. Secondary Outcome: GALAXI 1: Percentage of Participants With Clinical-Biomarker Response at Week 12
Time Frame: At Week 12
Reporting Status: Not Posted, anticipated posting 2031-06

14. Secondary Outcome: GALAXI 1: Percentage of Participants With Endoscopic Response at Week 12
Time Frame: At Week 12
Reporting Status: Not Posted, anticipated posting 2031-06

15. Secondary Outcome: Global: GALAXI 2 and 3: Percentage of Participants With Clinical Response at Week 4
Time Frame: At Week 4
Reporting Status: Not Posted, anticipated posting 2031-06

16. Secondary Outcome: Global: GALAXI 2 and 3: Percentage of Participants With Clinical Remission at Week 12
Time Frame: At Week 12
Reporting Status: Not Posted, anticipated posting 2031-06

17. Secondary Outcome: Global: GALAXI 2 and 3: Percentage of Participants With Endoscopic Response at Week 12
Time Frame: At Week 12
Reporting Status: Not Posted, anticipated posting 2031-06

18. Secondary Outcome: Global: GALAXI 2 and 3: Percentage of Participants With Fatigue Response at Week 12
Time Frame: At Week 12
Reporting Status: Not Posted, anticipated posting 2031-06

19. Secondary Outcome: Global: GALAXI 2 and 3: Percentage of Participants With Both Clinical Remission and Endoscopic Response at Week 12
Time Frame: At Week 12
Reporting Status: Not Posted, anticipated posting 2031-06

20. Secondary Outcome: Global: GALAXI 2 and 3: Percentage of Participants With Endoscopic Remission at Week 12
Time Frame: At Week 12
Reporting Status: Not Posted, anticipated posting 2031-06

21. Secondary Outcome: Global: GALAXI 2 and 3: Percentage of Participants With Both Clinical Response at Week 12 and Corticosteroid-Free Clinical Remission at Week 48
Time Frame: At Week 48
Reporting Status: Not Posted, anticipated posting 2031-06

22. Secondary Outcome: Global: GALAXI 2 and 3: Percentage of Participants With Both Clinical Response at Week 12 and Endoscopic Remission at Week 48
Time Frame: At Week 48
Reporting Status: Not Posted, anticipated posting 2031-06

23. Secondary Outcome: Global: GALAXI 2 and 3: Percentage of Participants With Clinical Remission at Week 48
Time Frame: At Week 48
Reporting Status: Not Posted, anticipated posting 2031-06

24. Secondary Outcome: Global: GALAXI 2 and 3: Percentage of Participants With Endoscopic Response at Week 48
Time Frame: At Week 48
Reporting Status: Not Posted, anticipated posting 2031-06

25. Secondary Outcome: Global: GALAXI 2 and 3: Percentage of Participants With Both Clinical Remission and Endoscopic Response at Week 48
Time Frame: At Week 48
Reporting Status: Not Posted, anticipated posting 2031-06

26. Secondary Outcome: Global: GALAXI 2 and 3: Percentage of Participants With Endoscopic Remission at Week 48
Time Frame: At Week 48
Reporting Status: Not Posted, anticipated posting 2031-06

27. Secondary Outcome: Global: GALAXI 2 and 3: Percentage of Participants With Deep Remission at Week 48
Time Frame: At Week 48
Reporting Status: Not Posted, anticipated posting 2031-06

28. Secondary Outcome: Regional: GALAXI 2 and 3: Percentage of Participants With PRO-2 Remission at Week 12
Time Frame: At Week 12
Reporting Status: Not Posted, anticipated posting 2031-06

29. Secondary Outcome: Regional: GALAXI 2 and 3: Percentage of Participants With Fatigue Response at Week 12
Time Frame: At Week 12
Reporting Status: Not Posted, anticipated posting 2031-06

30. Secondary Outcome: Regional: GALAXI 2 and 3: Percentage of Participants With Endoscopic Remission at Week 12
Time Frame: At Week 12
Reporting Status: Not Posted, anticipated posting 2031-06

31. Secondary Outcome: Regional: GALAXI 2 and 3: Percentage of Participants With Corticosteroid-free Clinical Remission at Week 48
Time Frame: At Week 48
Reporting Status: Not Posted, anticipated posting 2031-06

32. Secondary Outcome: Regional: GALAXI 2 and 3: Percentage of Participants With Endoscopic Response at Week 48
Time Frame: At Week 48
Reporting Status: Not Posted, anticipated posting 2031-06

33. Secondary Outcome: Regional: GALAXI 2 and 3: Percentage of Participants With Endoscopic Remission at Week 48
Time Frame: At Week 48
Reporting Status: Not Posted, anticipated posting 2031-06

34. Secondary Outcome: Regional: GALAXI 2 and 3: Percentage of Participants With Clinical Remission at Week 48
Time Frame: At Week 48
Reporting Status: Not Posted, anticipated posting 2031-06

35. Secondary Outcome: Regional: GALAXI 2 and 3: Percentage of Participants With Endoscopic Response at Week 48
Time Frame: At Week 48
Reporting Status: Not Posted, anticipated posting 2031-06

36. Secondary Outcome: Regional: GALAXI 2 and 3: Percentage of Participants With Durable Clinical Remission at Week 48
Time Frame: At Week 48
Reporting Status: Not Posted, anticipated posting 2031-06

37. Secondary Outcome: Regional: GALAXI 2 and 3: Percentage of Participants With PRO-2 Remission at Week 48
Time Frame: At Week 48
Reporting Status: Not Posted, anticipated posting 2031-06

38. Secondary Outcome: Regional: GALAXI 2 and 3: Percentage of Participants With Both Clinical Remission at Week 48 and Endoscopic Response at Week 48
Time Frame: At Week 48
Reporting Status: Not Posted, anticipated posting 2031-06

39. Secondary Outcome: Regional: GALAXI 2 and 3: Percentage of Participants With Corticosteroid-free Remission at Week 48
Time Frame: At Week 48
Reporting Status: Not Posted, anticipated posting 2031-06

ADVERSE EVENTS:
Time Frame: From Week 0 up to Week 48
Description: All Cause Mortality: All randomized participants. Serious adverse event (AE)/Other AEs: GALAXI 1: Safety analysis set: all participants who were randomized and received at least 1 dose of study intervention (including partial dose); GALAXI 2 and 3: All treated safety analysis set: all randomized participants who received at least 1 (partial or complete) dose of study intervention. GALAXI 1: MedDRA version (v)23.0, GALAXI 2 & 3:MedDRA v26.0. As planned, safety data was analyzed per intervention.
Groups:
- GALAXI 1 (Group 5) Placebo q4w; GALAXI 2 (Group 4) Placebo q4w; GALAXI 3 (Group 4) Placebo q4w: Participants randomized to receive placebo IV infusion q4w, excluding data after participant crossed over to ustekinumab.
- GALAXI 1 (Group 5) Placebo Followed by Ustekinumab 6 mg/kg IV Then 90 mg SC q8w; GALAXI 2 (Group 4) Placebo Followed by Ustekinumab 6 mg/kg IV Then 90 mg SC q8w; GALAXI 3 (Group 4) Placebo Followed by Ustekinumab 6 mg/kg IV Then 90 mg SC q8w: Participants randomized to receive placebo IV infusion q4w who crossed over to ustekinumab. Data in this group occurred after a participant crossed over to ustekinumab.
Arm/Group | GALAXI 1 (Group 1) Guselkumab 1200 mg IV q4w Followed by 200 mg SC q4w | GALAXI 1 (Group 2) Guselkumab 600 mg IV q4w Followed by 200 mg SC q4w | GALAXI 1 (Group 3) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w | GALAXI 1 (Group 4) Ustekinumab 6 mg/kg IV Followed by 90 mg SC q8w | GALAXI 1 (Group 5) Placebo q4w | GALAXI 1 (Group 5) Placebo Followed by Ustekinumab 6 mg/kg IV Then 90 mg SC q8w | GALAXI 2 (Group 1) Guselkumab 200 mg IV q4w Followed by 200 mg SC q4w | GALAXI 2 (Group 2) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w | GALAXI 2 (Group 3) Ustekinumab 6 mg/kg IV Followed by 90 mg SC q8w | GALAXI 2 (Group 4) Placebo q4w | GALAXI 2 (Group 4) Placebo Followed by Ustekinumab 6 mg/kg IV Then 90 mg SC q8w | GALAXI 3 (Group 1) Guselkumab 200 mg IV q4w Followed by 200 mg SC q4w | GALAXI 3 (Group 2) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w | GALAXI 3 (Group 3) Ustekinumab 6 mg/kg IV Followed by 90 mg SC q8w | GALAXI 3 (Group 4) Placebo q4w | GALAXI 3 (Group 4) Placebo Followed by Ustekinumab 6 mg/kg IV Then 90 mg SC q8w
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/73 | 0/73 | 0/71 | 0/70 | 0/43 | 0/148 | 0/149 | 0/150 | 0/77 | 0/49 | 0/151 | 0/148 | 0/150 | 0/76 | 0/51
Serious Adverse Events (participants affected / at risk) | 5/73 | 5/73 | 6/73 | 9/71 | 6/70 | 0/43 | 6/148 | 19/148 | 18/150 | 6/77 | 3/49 | 15/151 | 13/148 | 17/150 | 10/76 | 6/51
Other Adverse Events (participants affected / at risk) | 33/73 | 34/73 | 34/73 | 44/71 | 27/70 | 16/43 | 80/148 | 66/148 | 78/150 | 21/77 | 15/49 | 80/151 | 69/148 | 73/150 | 30/76 | 19/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GALAXI 1 (Group 1) Guselkumab 1200 mg IV q4w Followed by 200 mg SC q4w (N=73) | GALAXI 1 (Group 2) Guselkumab 600 mg IV q4w Followed by 200 mg SC q4w (N=73) | GALAXI 1 (Group 3) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w (N=73) | GALAXI 1 (Group 4) Ustekinumab 6 mg/kg IV Followed by 90 mg SC q8w (N=71) | GALAXI 1 (Group 5) Placebo q4w (N=70) | GALAXI 1 (Group 5) Placebo Followed by Ustekinumab 6 mg/kg IV Then 90 mg SC q8w (N=43) | GALAXI 2 (Group 1) Guselkumab 200 mg IV q4w Followed by 200 mg SC q4w (N=148) | GALAXI 2 (Group 2) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w (N=148) | GALAXI 2 (Group 3) Ustekinumab 6 mg/kg IV Followed by 90 mg SC q8w (N=150) | GALAXI 2 (Group 4) Placebo q4w (N=77) | GALAXI 2 (Group 4) Placebo Followed by Ustekinumab 6 mg/kg IV Then 90 mg SC q8w (N=49) | GALAXI 3 (Group 1) Guselkumab 200 mg IV q4w Followed by 200 mg SC q4w (N=151) | GALAXI 3 (Group 2) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w (N=148) | GALAXI 3 (Group 3) Ustekinumab 6 mg/kg IV Followed by 90 mg SC q8w (N=150) | GALAXI 3 (Group 4) Placebo q4w (N=76) | GALAXI 3 (Group 4) Placebo Followed by Ustekinumab 6 mg/kg IV Then 90 mg SC q8w (N=51)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angina Unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0
Anal Fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Aphthous Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Crohn's Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 5 | 3 | 3 | 1 | 3 | 4 | 1 | 6 | 2
Enterovesical Fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Frequent Bowel Movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal Tract Irritation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileal Stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Inflammatory Bowel Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 1
Intestinal Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Intestinal Stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Large Intestinal Stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0
Small Intestinal Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small Intestinal Stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bile Duct Stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatitis Toxic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abscess Intestinal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess Limb (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal Abscess (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacterial Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Covid-19 Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device Related Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis Infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal Fistula Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Liver Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post Procedural Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative Wound Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Testicular Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular Device Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural Intestinal Perforation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skull Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Liver Function Test Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Calcium Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis Enteropathic (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Desmoid Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Follicular Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal Tract Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wernicke's Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adjustment Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adjustment Disorder with Depressed Mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression Suicidal (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Calculus Urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine Polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Miscarriage of Partner (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GALAXI 1 (Group 1) Guselkumab 1200 mg IV q4w Followed by 200 mg SC q4w (N=73) | GALAXI 1 (Group 2) Guselkumab 600 mg IV q4w Followed by 200 mg SC q4w (N=73) | GALAXI 1 (Group 3) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w (N=73) | GALAXI 1 (Group 4) Ustekinumab 6 mg/kg IV Followed by 90 mg SC q8w (N=71) | GALAXI 1 (Group 5) Placebo q4w (N=70) | GALAXI 1 (Group 5) Placebo Followed by Ustekinumab 6 mg/kg IV Then 90 mg SC q8w (N=43) | GALAXI 2 (Group 1) Guselkumab 200 mg IV q4w Followed by 200 mg SC q4w (N=148) | GALAXI 2 (Group 2) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w (N=148) | GALAXI 2 (Group 3) Ustekinumab 6 mg/kg IV Followed by 90 mg SC q8w (N=150) | GALAXI 2 (Group 4) Placebo q4w (N=77) | GALAXI 2 (Group 4) Placebo Followed by Ustekinumab 6 mg/kg IV Then 90 mg SC q8w (N=49) | GALAXI 3 (Group 1) Guselkumab 200 mg IV q4w Followed by 200 mg SC q4w (N=151) | GALAXI 3 (Group 2) Guselkumab 200 mg IV q4w Followed by 100 mg SC q8w (N=148) | GALAXI 3 (Group 3) Ustekinumab 6 mg/kg IV Followed by 90 mg SC q8w (N=150) | GALAXI 3 (Group 4) Placebo q4w (N=76) | GALAXI 3 (Group 4) Placebo Followed by Ustekinumab 6 mg/kg IV Then 90 mg SC q8w (N=51)
Anaemia (Blood and lymphatic system disorders) | 3 | 6 | 1 | 7 | 4 | 1 | 10 | 8 | 11 | 3 | 1 | 5 | 7 | 5 | 5 | 3
Abdominal Pain (Gastrointestinal disorders) | 2 | 2 | 1 | 5 | 3 | 0 | 9 | 11 | 13 | 3 | 1 | 5 | 8 | 12 | 4 | 0
Crohn's Disease (Gastrointestinal disorders) | 4 | 5 | 6 | 11 | 4 | 5 | 12 | 8 | 12 | 8 | 2 | 11 | 10 | 11 | 8 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 4 | 2 | 2 | 0 | 5 | 6 | 3 | 0 | 1 | 3 | 3 | 11 | 3 | 1
Nausea (Gastrointestinal disorders) | 2 | 2 | 3 | 4 | 2 | 0 | 5 | 5 | 6 | 1 | 0 | 4 | 4 | 4 | 6 | 0
Pyrexia (General disorders) | 4 | 3 | 6 | 5 | 2 | 1 | 8 | 10 | 14 | 5 | 1 | 8 | 9 | 12 | 3 | 3
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 22 | 18 | 24 | 2 | 7 | 31 | 27 | 16 | 8 | 5
Nasopharyngitis (Infections and infestations) | 8 | 9 | 8 | 8 | 3 | 4 | 10 | 7 | 12 | 2 | 1 | 11 | 5 | 7 | 3 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 6 | 2 | 7 | 6 | 2 | 12 | 15 | 10 | 3 | 2 | 13 | 14 | 13 | 3 | 5
Alanine Aminotransferase Increased (Investigations) | 2 | 1 | 5 | 0 | 1 | 1 | 2 | 1 | 2 | 0 | 1 | 5 | 1 | 0 | 1 | 0
Haemoglobin Decreased (Investigations) | 3 | 2 | 1 | 1 | 5 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 8 | 5 | 4 | 3 | 14 | 14 | 12 | 4 | 3 | 11 | 9 | 8 | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 3 | 2 | 0 | 1 | 6 | 5 | 3 | 2 | 0 | 4 | 3 | 0 | 1 | 0
Headache (Nervous system disorders) | 7 | 10 | 5 | 6 | 1 | 4 | 16 | 6 | 13 | 3 | 1 | 8 | 9 | 6 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT03466411/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT03466411/SAP_001.pdf